CLINICAL TRIAL: NCT00834483
Title: Use of Knotless Suture for Closure of Total Hip and Knee Arthroplasties: A Prospective-randomized Clinical Trial
Brief Title: Use of Knotless Suture for Closure of Total Hip and Knee Arthroplasties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brett Levine, MD, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08091607
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
Keywords: Safety; Efficacy; Cost-savings; Cosmesis; Safety and efficacy of wound closure; Cost-savings potential; Cosmesis of the wound/scar
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Knotless suture for wound closure
  Interventions: Device: Knotless suture for wound closure
- 2 (Active Comparator): Layered traditional wound closure (monocryl)
  Interventions: Device: Layered traditional wound closure (monocryl)

INTERVENTIONS:
Device: Knotless suture for wound closure — Angiotech Quill SRS
  Other Names: Angiotech Quill SRS
  Arms: 1
Device: Layered traditional wound closure (monocryl) — Layered traditional wound closure (monocryl)
  Other Names: Monocryl
  Arms: 2

SUMMARY:
Barbed sutures offer several potential advantages in layered wound closure of hip and knee replacement surgeries. It use is gaining increased acceptance across many of the other surgical disciplines at this time. The purpose of this study is to evaluate the use of Quill as part of our layered closure compared to using our traditional sutures. The study timeline begins at the time of the surgical procedure and continues through the routine follow-up of total joint replacements at 2, 6, and 12 weeks, and will conclude at the six month post-operative office visit.

Primary Objectives:

* To evaluate the safety and efficacy of wound closure in primary hip and knee replacements using a bidirectional barbed suture (knotless) compared to a traditional layered (vicryl) wound closure.

Secondary Objectives:

* Establish the all around (intra-operative and post-operative) cost-savings potential in using a knotless wound closure compared to that of a layered vicryl closure (our standard suture protocol).
* Assess the overall cosmesis of the wound/scar as well as perceived presence of subcutaneous surgical knots, when using the knotless wound closure versus our traditional layered suture closure.

DETAILED DESCRIPTION:
We performed a prospective, randomized clinical trial to evaluate the efficacy of using a bidirectional barbed suture compared with traditional sutures in the deep closure of primary total hip (25) and knee (35) arthroplasties. Complications, time to closure, and length of surgery were evaluated. Closure was noted to be significantly faster (9.3 vs 13.6 minutes, P b .005) in the barbed suture group. Wound-related complications were similar (3 cases) in both groups at 3-month follow-up. Although this study supports the use of barbed technology as a functionally comparable and more efficient modality of wound closure with the potential for costs savings based on reduced operative time, the cost-effectiveness of its adoption is institution dependent and will rely on the optimization of all other perioperative factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female of any race
* Ages 18-80 years old
* Patients must be undergoing a primary hip or knee arthroplasty
* Patients must be able to understand and willing to cooperate with study procedures
* Able to provide written and verbal informed consent

Exclusion Criteria:

* Allergy or intolerance to the study materials
* Surgical intervention during the past month for the treatment of the painful joint or its underlying etiology
* History of previous surgeries on the affected joint other than arthroscopy (open surgeries)
* History of any substance abuse or dependence within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett R Levine, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush university Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Greenberg JA, Einarsson JI. The use of bidirectional barbed suture in laparoscopic myomectomy and total laparoscopic hysterectomy. J Minim Invasive Gynecol. 2008 Sep-Oct;15(5):621-3. doi: 10.1016/j.jmig.2008.06.004. Epub 2008 Jul 10. PMID 18619922
- [Background] Moran ME, Marsh C, Perrotti M. Bidirectional-barbed sutured knotless running anastomosis v classic Van Velthoven suturing in a model system. J Endourol. 2007 Oct;21(10):1175-8. doi: 10.1089/end.2007.9913. PMID 17949320
- [Background] Villa MT, White LE, Alam M, Yoo SS, Walton RL. Barbed sutures: a review of the literature. Plast Reconstr Surg. 2008 Mar;121(3):102e-108e. doi: 10.1097/01.prs.0000299452.24743.65. PMID 18317092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-blinded, prospective, randomized trial was conducted from February 2009 through June 2009 and was approved by our institutional review board. Recruitment was in our office only.
Pre-assignment Details: No participants were excluded except those that would not sign consent. 5 patients were excluded as they did not want to participate giving us 65 offers and 60 enrollments.
Groups:
- Treatment Group: Knotless suture for wound closure
- Control Group: Layered traditional wound closure (monocryl)
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.86) | 63.5 (10.8) | 63.95 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Closure Time
Description: We performed a prospective, randomized clinical trial to evaluate the efficacy of using a bidirectional barbed suture compared with traditional sutures in the deep closure of primary total hip (25) and knee (35) arthroplasties. Complications, time to closure, and length of surgery were evaluated.
Time Frame: 6 months
Population: A power analysis was performed based on mean closure times by the 2 surgeons and determined that a sample size of 23 patients in each group would provide 90% power to detect a 50% difference in closure time. To account for patients being lost to FU, we enrolled 29 to the traditional closure group and 31 to the barbed closure group
Measure: Mean (Full Range); unit: Average time in minutes
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 31 | 29
Average time in minutes | 9.34 [5.4 to 13.8] | 13.57 [7.0 to 26.2]

2. Secondary Outcome: Cost-analysis
Description: Cost savings included the material costs and then we factored in the time savings in the OR. The OR time was based upon the average cost per minute to work in one of our ORs
Time Frame: 1 year
Population: Power analysis was performed as above.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 31 | 29
Dollars | 52.75 (19.96) | 12.79 (1.95)

3. Secondary Outcome: Visual Analog Score, Cosmesis
Description: Overall cosemesis was graded by patient and surgeon. This is based on a 1-6 scale, with a 6 being a perfect score based upon satisfaction with the wound cosmesis.
  1 is an unacceptable or poor perspective in regards to wound cosmesis.
Time Frame: 6 months
Population: Power analysis described above
Measure: Mean (Full Range); unit: units on a scale (1 is a low score)
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 31 | 29
units on a scale (1 is a low score) | 5.9 [1 to 6] | 5.8 [1 to 6]

ADVERSE EVENTS:
Arm/Group | Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/29
Other Adverse Events (participants affected / at risk) | 2/31 | 3/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=31) | Control Group (N=29)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient fell after surgery. Not related to the treatment arm, but required re-operation for arthrotomy rupture.
OTHER ADVERSE EVENTS (reported when occurring in more than 3.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=31) | Control Group (N=29)
incisional erythema (Infections and infestations) | 2 (2) | 3 (3) — 2 in the barbed suture and 3 in the traditional closure group developed incisional erythema, and all resolved with oral antibiotics.

LIMITATIONS AND CAVEATS:
Five patients were offered enrollment but refused to participate, however this does not alter our data as sixty others did enroll.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No